CLINICAL TRIAL: NCT02120326
Title: Randomised Double-blind Evaluation of the Prophylactic Efficacy of Transcranial Direct Current Stimulation (tDCS) in Chronic Migraine
Brief Title: Evaluation of the Prophylactic Efficacy of tDCS in Chronic Migraine
Acronym: Medis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DCIC13/48
Record Dates: First submitted 2014-04-15; First posted 2014-04-22 (Estimated); Last update posted 2025-08-13 (Actual); Status verified 2020-11

CONDITIONS: Chronic Migraine as Defined by Criteria of International Headache Society (IHS)
Keywords: Chronic migraine, tDCS, Transcranial direct current stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- active tDCS (Experimental)
  Interventions: Device: Transcranial direct current stimulation of the motor cortex
- simulated tDCS (Placebo Comparator)
  Interventions: Device: simulation of Transcranial direct current stimulation of the motor cortex

INTERVENTIONS:
Device: Transcranial direct current stimulation of the motor cortex — The area of stimulation is determined by by EEG system 10/20. The two electrodes are soaked in saline and then placed on the scalp.
  Stimulation parameters:
  * 2 mA intensity
  * Continuous stimulation for 20 min with rise times and fall times of 10 seconds each
  Arms: active tDCS
Device: simulation of Transcranial direct current stimulation of the motor cortex — The area of stimulation is determined by by EEG system 10/20. The two electrodes are soaked in saline and then placed on the scalp.
  Stimulation parameters:
  * The intensity of the stimulation current is 2 mA
  * The current is applied during the first 30 seconds with rise times and fall times of 10 seconds each. Then the session will be continued without actual stimulation.
  Arms: simulated tDCS

SUMMARY:
The purpose of this study is to determine whether TDCS is an effective prophylactic therapy of chronic migraine.

DETAILED DESCRIPTION:
Consenting patients will report on a book, all of their migraine attack for 1 month. Then they will be randomized to the active tDCS group or sham tDCS group. Patients will have one session of tDCS per day during the first week, then one session per week for a month and finally a session every 15 days for 1 month. After tDCS sessions, patients will be followed for 3 months. Throughout their participation in the study, patients will complete their migraine record (1month of base line before tDCS, 2 months during tDCS, 3 months after tDCS).

Patients will have 5 evaluation examinations:

* The first, one before tDCS,
* The second, 1 month after the beginning of tDCS
* The third, immediately after the end of tDCS
* The fourth, 1 month after the end of tDCS
* And the last one, 3 months after the end of tDCS.

The physician responsible for conducting tDCS sessions will make the randomization via a website.

The physician in charge of the evaluation examinations will don't know the allocated treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic migraine for more than 1 year
* Stable treatment since 1 month
* Frequency of migraine crisis is above 8 per month during last month
* chronic migraine that has not been improved over the previous year by at least 3 different prophylactic treatments recommended and well conducted
* Patient agreeing not to try other migraine prophylactic treatment, throughout the study
* Patient's written consent

Exclusion Criteria:

* History of drug addiction, epilepsy, or severe head trauma with bone break
* History of psychiatric illness (psychosis and severe cognitive disorders) may interfere with the proper conduct of the study
* Presence of intracranial ferromagnetic material or an implanted stimulator
* Introduction of a new treatment for less than a month
* Pregnant women, parturient women, breast-feeding mother. Lack of effective contraception
* Person not understanding the study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-05-05 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2020-06-23 (Actual)

PRIMARY OUTCOMES:
Comparison of the evolution of seizure frequency between the two groups | Evolution of seizure frequency since base line to 3 months after the end of tDCS

SECONDARY OUTCOMES:
Comparison of the evolution of seizure severity between the two groups | Evolution of seizure severity since base line to 3 months after the end of tDCS
  Headache Impact Test 6 (HIT-6) questionnaire
Comparison of the evolution of crisis treatment use between the two groups | Evolution of crisis treatment use since base line until 3 months after the end of tDCS
  Frequency of taking crisis treatment. After each crisis, taking crisis treatment will be noted by the patient on his migraine record book.
Comparison of the evolution of the disease impact between the two groups | Evolution of the disease impact since base line to 3 months after the end of tDCS
  Migraine Disability Assessment Scale (MIDAS) scale
Comparison of the evolution of the patient satisfaction between the two groups | Evolution of the patient satisfaction since base line to 3 months after the end of tDCS
  Clinical Global Impression (CGI) scale
Comparison of the evolution of the quality of life between the two groups | Evolution of the quality of life since base line until 3 months after the end of tDCS
  Short Form 12 (SF-12) quality of life questionnaire
Comparison of the evolution of anxiety and depression levels between the two groups | Evolution of anxiety and depression levels since base line until 3 months after the end of tDCS
  Hospital Anxiety and Depression scale (HAD) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: HODAJ Hasan, MD, Principal Investigator — University Hospital, Grenoble
Locations (2):
- France (2):
  - Grenoble University Hospital, Grenoble, Isere
  - Hospital of Voiron, Voiron, Isere

REFERENCES:
- [Result] Hodaj H, Payen JF, Mick G, Vercueil L, Hodaj E, Dumolard A, Noelle B, Delon-Martin C, Lefaucheur JP. Long-term prophylactic efficacy of transcranial direct current stimulation in chronic migraine. A randomised, patient-assessor blinded, sham-controlled trial. Brain Stimul. 2022 Mar-Apr;15(2):441-453. doi: 10.1016/j.brs.2022.02.012. Epub 2022 Feb 25. PMID 35219923